CLINICAL TRIAL: NCT05102448
Title: Comparison of the Efficacy and Safety of Tofacitinib and Methotrexate Based on Prednisone Therapy in Patients with Active Phase of Takayasu's Arteritis: a Randomized Controlled Trial
Brief Title: Comparison of Tofacitinib and Methotrexate in Takayasu's Arteritis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Jiang lindi, Ph.D, M.D., Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TACTIC-TM
Record Dates: First submitted 2021-10-19; First posted 2021-11-01 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Takayasu Arteritis
MeSH Terms: conditions — Takayasu Arteritis | interventions — tofacitinib; Methotrexate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tofacitinib (Experimental): Partcipants would be given one tablet of tofacitinib (5mg per tablet), twice per day, the treatment duration will last 12 months during the whole follow-up period.
  Interventions: Drug: Tofacitinib
- Methotrexate (Active Comparator): Participates would be given tablets of methotrexate (2.5mg per tablet) 15mg each week, the treatment duration will last 12 months during the whole follow-up period.
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Tofacitinib — 1. Tofacitinib 5mg twice a day for 12 months;
  2. Basic treatment with prednisone: (1) the initial dose of prednisone (or equivalent): 0.8mg/kg/day (maximum 60mg/day). (2) Glucocorticoids tapering: glucocorticoids is tapered after two weeks treatment and is tapered 5mg each 2 weeks to 10mg qd in the first 6 months if patients were in inactive status based on the NIH disease activity criteria. During the 6th to 12th month, glucocorticoids is tapered 2.5mg each 4 weeks until 7.5mg qd if patients were in inactive status based on the NIH disease activity criteria.
  Other Names: TOF
  Arms: Tofacitinib
Drug: Methotrexate — 1. Methotrexate (15mg each week) for 12 months
  2. Basic treatment with prednisone: (1) the initial dose of prednisone (or equivalent): 0.8mg/kg/day (maximum 60mg/day). (2) Glucocorticoids tapering: glucocorticoids is tapered after two weeks treatment and is tapered 5mg each 2 weeks to 10mg qd in the first 6 months if patients were in inactive status based on the NIH disease activity criteria. During the 6th to 12th month, glucocorticoids is tapered 2.5mg each 4 weeks until 7.5mg qd if patients were in inactive status based on the NIH disease activity criteria.
  Other Names: MTX
  Arms: Methotrexate

SUMMARY:
The aim of this study is to evaluate and compare the efficacy and safety of tofacitinib and methotrexate based on prednisone therapy in patients with Takayasu arteritis

DETAILED DESCRIPTION:
Takayasu's arteritis (TAK), a chronic large vessel vasculitis, involves the aorta and its main branches. Glucocorticoids and immunosuppressants such as methotrexate, cyclophosphamide are common agents for TAK treatment. However, their effects for remission induction and relapse prevention are not satisfied. More effective agents for TAK treatment remain to be investigated. Tofacitinib (TOF) is a Jak inhibitor, which has been proved to be effective in multiple autoimmune diseases such as rheumatoid arthritis. Our preliminary real-world study also demonstrated a promising treatment effect of TOF in patients with TAK. But its efficacy and safety needs further verification. The present randomized controlled trial aimes to compare efficacy between methotrexate and tofacitinib in TAK treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients met 1990 American College of Rheumatology (ACR) classification criteria or 2018 ACR classification criteria (draft) of TAK
2. Women or men aged 18-65
3. All patients agreed that there is no fertility plan during clinical trials, and the results of female serum or urinary pregnancy tests must be negative
4. Active TAK patients according to NIH disease activity criteria
5. All patients agreed to sign the informed consent

Exclusion Criteria:

1. Patients with organ failure who accord to one or more of the following conditions:

   I.Heart function New York class 4 II.Glomerular filtration rate ≤ 60ml/min III.Liver function Child grade 2 and above IV.High-frequency melanoma (attacks for 3 consecutive days) V.Acute cerebral infarction or cerebral hemorrhage VI.Blood pressure > 160/100mmHg
2. Patients who received revascularization surgery related to the treatment of TAK within 3 months (except balloon dilatation); balloon dilatation or surgery unrelated to TAK within 1 month
3. Patients who have other autoimmune diseases (e.g. ANCA-associated vasculitis, systemic lupus erythematosus, Behcet's disease, etc.)
4. Patients with severe, progressive or uncontrolled comorbidities of kidney, liver, blood system, gastrointestinal, lung, heart, etc or other coexisting medical conditions that may exert unexpected risks
5. Patients with concomitant diseases, such as asthma, that may require additional medium to high doses of glucocorticoids (prednisone ≥ 10mg/ days or equivalent dose) during the study period
6. Patients with active infections with HBV, HCV, tuberculosis or other serious acute or chronic infections
7. Patients with malignancies
8. Patients with one or more of the following abnormal laboratory examinations I.Serum ALT or AST ≥ 1.5 times the normal upper limit; II.White blood cell count ≤ 4 × 109/L III.Platelet count ≤ 100x109/L IV.Hemoglobin < 85g/L V.Other abnormal laboratory tests that may cause unacceptable risks
9. Patients allergic to the experimental drug
10. Patients who have ever failed to tofacitinib or methotrexate after 3 months' treatment in previous medical history

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The effectiveness rate after 6 months' treatment | From the enrollment to the end of 6 months
  The effectiveness rate equals to patients who achieved this goal /patients at the end of 6 months. The effectiveness was defined as satisfying three of the following 1)-4) criteria and the 5) criteria: 1) no systemic symptoms such as weakness, weight loss, etc; 2) no new ischemic symptoms or signs; 3) normal erythrocyte sedimentation rate (ESR); 4) no new vascular progression or new lesions upon imaging; 5) GCs is tapered to 10mg qd and this dosage is maintained for 4 weeks.

SECONDARY OUTCOMES:
The remission rate with GCs 7.5mg qd at the end of 12 months | From the enrollment to the the end of 12 months
  Ratio of patients who achieved remission with GCs 7.5mg qd at the end of 12 months. The remission is defined as satisfying three of the following 1)-4) criteria: 1) no systemic symptoms such as weakness, weight loss, etc; 2) no new ischemic symptoms or signs; 3) normal erythrocyte sedimentation rate (ESR); 4) no new vascular progression or new lesions upon imaging. It is required that GCs 7.5mg qd should be maintained at least for four weeks.
Relapse free survival rate | From the enrollment to the the end of 12 month
  Ratio of patients without relapse after achieving remission during the 12 months follow-up
The cumulative dosage of GCs during the whole period of 12-months follow-up | From the enrollment to the the end of 12 months
  The cumulative dosage = Sum of doses of prednisone （or equivalents） each day
Side effects rate | From the enrollment to the the end of 12 months
  Ratio of patients with side effects. All the kinds of adverse event related to the treatment and the disease itself will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Lindi Jiang, Ph.D., M.D., Study Chair — Department of Rheumatology in Zhongshan hospital, Fudan University
Locations (1):
- Lindi Jiang, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No